CLINICAL TRIAL: NCT06057311
Title: Effectiveness of Equine Assisted Therapy in Children With Autism Spectrum Disorder: A Randomized Controlled Study
Brief Title: Equine Assisted Therapy in Autism Spectrum Disorder
Acronym: AUTISM-EAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Collaborators: Turkey Jockey Club Equine Therapy Center, Izmir, Turkey (Unknown)
Responsible Party: Principal Investigator, Betül Taşpınar, Principal Investigator, Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AUTISM-EAT-35
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Equine-Assisted Therapy; Autism Spectrum Disorder
Keywords: Equine-assisted therapy; Hippotherapy; Autism spectrum disorder; Sleep; Balance; Activities of daily living; Quality of life
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hippotherapy Group (Experimental): The sessions for the HTG were conducted on horseback by a "leader", "side walker", and "physiotherapist" while the child was mounted on the horse. Before mounting, the child was dressed in the safety equipment of a helmet and rider vest by the physiotherapist and was directed to mount the horse from the mounting steps. In the first week of training, the cases received adaptation training. Within the training, 7 min of simple sitting on the horse were performed. In this position, the child was able to caress the horse's neck with one or both hands, rest while the horse walked, and 10 standing (or for those who could not do this, the horse was in a standing position)n the stirrups exercises were performed while holding the retaining strap.
  Interventions: Other: Hippotherapy
- Equine-Assisted Activities Therapy Group (Experimental): Under the guidance of the physiotherapist, the children in the EAATG performed routine care of the horse, such as grooming, feeding, and hoof care. During equine-assisted activities, the physiotherapist ensured the correct positioning of the child's body when approaching the horse using equipment and during movement. The study participants groomed the horse, wiped the horse's feathers with a towel, combed the mane, checked the hooves, cleaned out any grit, and performed the procedures for the horse to go out. Finally, the child gave food and water to the horse, said farewell and left the therapy area.
  Interventions: Other: Equine-Assisted Activities Therapy
- Control Group (Other): The children in the control group were evaluated at the same time as the other groups but were not included in any therapy. All assessments were conducted at baseline and 6 weeks later. When the study was completed, the subjects in this group were permitted 10 sessions of hippotherapy if they so wished.
  Interventions: Other: Control

INTERVENTIONS:
Other: Hippotherapy — The participants in HT Group; received 12 sessions as 2 sessions a week for 6 weeks. Each therapy session lasted for an average of 20 min. The assessments were applied twice to all participants before and after the training. The treatments and assessments were performed by the same physiotherapist in the same environment.
  Other Names: HT
  Arms: Hippotherapy Group
Other: Equine-Assisted Activities Therapy — The participants in the EAAT Group received 12 sessions as 2 sessions a week for 6 weeks. Each therapy session lasted for an average of 20 min. The assessments were applied twice to all participants before and after the training. The treatments and assessments were performed by the same physiotherapist in the same environment.
  Other Names: EAAT
  Arms: Equine-Assisted Activities Therapy Group
Other: Control — The Control Group (CG) did not receive any training. The assessments were applied twice to CG at baseline and after 6 weeks. The treatments and assessments were performed by the same physiotherapist in the same environment.
  Arms: Control Group

SUMMARY:
Autism Spectrum Disorder (ASD) is a common neurodevelopmental disorder that negatively affects social interaction, communication, and behavior. Various animals have started to be used for therapeutic purposes by those in need. In recent years, especially equine-assisted therapies have become popular. However, it has been reported in the literature that more studies on this subject are needed. Therefore, the aim of this study was to examine the effects of equine-assisted therapy for children with autism on daily living activities, balance, quality of life, and sleep.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) was first defined by Leo Kanner in 1943 as a common neurodevelopmental disorder that has a negative effect on social interaction, communication, and behaviour. These individuals have problems such as impaired sensory processing skills, reduced balance and coordination, difficulties in undertaking daily living activities, diminished quality of life, sleep problems, and poor speech and language skills. According to the 2015 report published by the American National Autism Center, treatments are examined under three headings: those based on science, those promising, and those not based on science. Animal support therapies are included in the intervention not based on science.

It can be seen in the literature that the relationship between people and animals provides people with physical, mental and psychological support. Because of the positive effects of this relationship, various animals have started to be used for therapeutic purposes by those in need. Horses are used most often because accessibility is easy and they share many characteristics with humans. Therapies that include horses come under the following five headings: Adaptive Riding, Equine Assisted Activities, Equine Assisted Psychotherapy, Equine Assisted Therapy, and Hippotherapy.

Equine-assisted therapy is used in several pathologies and various age groups, most commonly in pediatric rehabilitation. However, there are few studies in the literature on this subject. Therefore, the aim of this study was to examine the effects of equine-assisted therapy for children with autism on daily living activities, balance, quality of life, and sleep. Thus, it is thought to contribute to the literature in terms of the effectiveness of applying equine-assisted therapies together with traditional therapies in individuals with autism spectrum disorder.

Study Hypothesis as follows: Equine-Assisted Therapies have an effect on daily living activities, balance, quality of life, and sleep of individuals with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ASD,
* Having <60 kg in body weight
* Having no shunt,
* Having no allergy to feathers or dust,
* Having not previously received equine-assisted therapy.

Exclusion Criteria:

* Having hip or shoulder dislocation, osteoporosis/coxarthrosis,
* Having uncontrollable seizures,
* Having aneurysm,
* Having a recent history of fracture,
* Having decubitus,
* Having atlantoaxial instability,
* Having hemophilia,
* Using anticoagulant drugs,
* Having acute arthritis,
* Having an unstable spine,
* Having acute disc hernia,
* Having spondylolisthesis,
* Having spinal fusion,
* Having no control of the head.

Other exclusion criteria related to therapies;

* Inability to adapt to the therapy,
* Having a fear of horses,
* The occurrence of seizures or worsening of the existing seizure status,
* Worsening of vital signs,
* Requesting to quit the study participation

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Assessment of Activities of Daily Living | Change from baseline at 6 weeks
  Activities of daily living (ADL) were evaluated with the Waisman Activities of Daily Living Scale (W-ADLS), for which validity and reliability studies were conducted in Turkey in 2016. The scale consists of 17 items scored from 0 (cannot do this at all) to 2 (can do this independently). The scale has higher points showing independence.
The Assessment of Balance | Change from baseline at 6 weeks
  The Paediatric Balance Scale (PBS) developed by Franjoine was used to evaluate balance. Validity and reliability studies of the scale in Turkish were conducted by Karali. The scale consists of 14 items evaluating daily activities of the child at home, school, and in the community. Each item is scored from 0 (the activity cannon be performed independently) to 4 (the activity is performed independently) giving a total score in the range of 0 - 56. Higher points indicate good balance.
Assessment of Quality of Life | Change from baseline at 6 weeks
  The original German healthy quality of life questionnaire (KINDL) was tested for validity and reliability in Turkish by Eser et al. in 2008. There are family forms (Kiddy Kindl Parents and Kid and Kiddo Kindl Parents) for children in the age ranges of 4 - 7 years and 8 - 12 years, who will not be able to complete the form. The family form of this questionnaire was used in this study. Total points range from 0 to 100, with higher points showing a good quality of life.
Assessment of Sleep Habits | Change from baseline at 6 weeks
  The sleep habits of the participants were evaluated using the short Turkish version of the Children's Sleep Habits Questionnaire (CSHQ), which was developed to assess the sleep habits and problems of children. The questionnaire consists of 33 items. The total score of the items is seen as 41 lines, and as the score increases, sleep habits change at a better rate. Turkish validity and reliability studies were conducted by Fis et al. in 2010.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Taspinar, Prof. Dr., Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No